CLINICAL TRIAL: NCT00197431
Title: Pharmacokinetic and Pharmacodynamic Study of S-1 and Its Effects in Patients With the Digestive Organ Cancer With Reference to Genetic Polymorphism and Activity of CYP2A6 and DPD
Brief Title: Pharmacokinetic and Pharmacodynamic Study of S-1 in Patients With Digestive Organ Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamamatsu University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-12005
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-03-22 (Estimated); Status verified 2003-12

CONDITIONS: Gastric Cancer; Esophageal Cancer; Pancreatic Cancer; Colon Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms | interventions — S 1 (combination)

INTERVENTIONS:
Drug: S-1

SUMMARY:
S-1 is a novel oral fluorouracil antitumor drug that consists of tegafur which is a prodrug of 5-fluorouracil (5-FU); 5-chloro-2,4-dihydropyridine (CDHP), which inhibits dihydropyrimidine dehydrogenase (DPD) activity; and potassium oxonate (Oxo), which reduces gastrointestinal toxicity. 5-FU is metabolized by CYP2A6 and DPD. In this study, the researchers investigate the influences of differences in activities of CYP2A6 and DPD on pharmacokinetics and pharmacodynamics of S-1 and clinical outcomes in digestive organ cancer patients treated with S-1.

ELIGIBILITY:
Inclusion Criteria:

* Patients with digestive organ cancer

Exclusion Criteria:

* Patients without digestive organ cancer

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-01

PRIMARY OUTCOMES:
Whether the differences in activities of CYP2A6 and DPD affect pharmacokinetics and pharmacodynamics of S-1 and clinical outcomes

SECONDARY OUTCOMES:
Side effect and motility of patients treated with S-1

CONTACTS AND LOCATIONS:
Overall Officials: Naohito Shirai, MD., PhD, Study Chair — Department Laboratory Medicine, Hamamatsu University School of Medicine
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Shizuoka, Japan